CLINICAL TRIAL: NCT05358912
Title: Does Targeted Abdominal Perfusion Pressure Reduce Renal Injury and Mortality in Septic Shock Patients? A Prospective Controlled Trial
Brief Title: Efficacy of Targeted Abdominal Perfusion Pressure in Septic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Uğur Bilgin, MD, Anesthesiology Specialist, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AbdominalPressure
Record Dates: First submitted 2022-04-18; First posted 2022-05-03 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Septic Shock; Septicemia; Intraabdominal Hypertension; Renal Injury
MeSH Terms: conditions — Shock, Septic; Sepsis; Intra-Abdominal Hypertension | interventions — Vasoconstrictor Agents; Crystalloid Solutions; Weights and Measures; Arterial Pressure

STUDY DESIGN:
Intervention Model Description: Patients in different groups will be subjected to different monitoring protocols.
  All will be treated according to designated target values.
Who Masked: Participant
Masking Description: Patients will be blind to their designated groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Patients who are diagnosed with septic shock and who have intra-abdominal pressure of less than 8 mmHg.
  Target mean arterial pressure is 65 mmHg and above.
  Interventions: Drug: Vasopressor Agent; Drug: Crystalloid Solutions; Procedure: Invasive Blood Pressure Monitoring; Procedure: Intra-Abdominal Pressure Monitoring
- MAP Group (Active Comparator): Patients who are diagnosed with septic shock and who have intra-abdominal pressure greater than 8 mmHg.
  Target mean arterial pressure is 65 mmHg and above.
  Interventions: Drug: Vasopressor Agent; Drug: Crystalloid Solutions; Procedure: Invasive Blood Pressure Monitoring; Procedure: Intra-Abdominal Pressure Monitoring
- APP Group (Experimental): Patients who are diagnosed with septic shock and who have intra-abdominal pressure greater than 8 mmHg.
  Target abdominal perfusion pressure is 65 mmHg and above.
  Interventions: Drug: Vasopressor Agent; Drug: Crystalloid Solutions; Procedure: Invasive Blood Pressure Monitoring; Procedure: Intra-Abdominal Pressure Monitoring; Other: Abdominal Perfusion Pressure

INTERVENTIONS:
Drug: Vasopressor Agent — Patients will receive vasopressor agents according to "Surviving Sepsis Campaign Guidelines 2021"
Drug: Crystalloid Solutions — Patients will receive crystalloid solutions according to "Surviving Sepsis Campaign Guidelines 2021"
Procedure: Invasive Blood Pressure Monitoring — Invasive blood pressure monitoring will be performed through an intra-arterial cannula placed in the radial artery. Philips Intellivue mx 500 monitors will be used for bedside monitoring.
  Other Names: Measurement for Mean Arterial Pressure
Procedure: Intra-Abdominal Pressure Monitoring — IAP will be measured indirectly by monitoring the pressure in the bladder.
  Bladder pressure will be measured through an indwelling Foley catheter every twelve hours. Twenty-five mL of sterile normal saline will be injected in each measurement and readings will be recorded with a pressure transducer.
Other: Abdominal Perfusion Pressure — APP will be calculated with the following formula: (Mean arterial pressure) - (Intra-abdominal Pressure)
  Arms: APP Group

SUMMARY:
Septic shock is a clinical condition that is defined as a subset of sepsis that causes very high mortality and morbidity.

Surviving sepsis campaign guideline states that the target mean arterial pressure should be 65 mmHg and above in septic shock patients. It is known that abdominal pressure increases and perfusion of intra-abdominal organs decreases in septic shock patients.

With this study, we aim to investigate the effects of targeted abdominal perfusion pressure (60 mmHg and above) on renal injury, reversal of renal injury, liver functions and ultimately mortality in patients with septic shock.

DETAILED DESCRIPTION:
Patients diagnosed with septic shock according to "Surviving Sepsis Campaign Guidelines 2021" will be included in the study.

Groups will be formed after the measurement of intra-abdominal pressure (IAP). Those with IAP of less than 8 mmHg will be assigned to the control group and treated according to mean arterial pressure. Those with IAP greater than 8 mmHg will be divided into two groups by computer-generated randomization (via randomizer.org). One group (Group MAP) will be treated according to mean arterial pressure and the other group (Group APP) will be treated according to abdominal perfusion pressure. In Group APP, maximum arterial pressure will be targeted as 130/85 mmHg.

All patients will receive appropriate antibiotic therapy, fluid therapy and, vasopressor treatment as recommended in "Surviving Sepsis Campaign Guidelines 2021" and abdominal pressure measurement will be repeated every 12 hours.

Age, sex, body mass index, cause of sepsis and comorbidities of all patients will be recorded.

Patients will be followed for liver and kidney function tests, procalcitonin and lactate levels, daily SOFA (Sequential Organ Failure Assessment) calculations, length of stay (days), length of stay in mechanical ventilator (days), and 30 and 90 days mortality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of septicemia according to "Surviving Sepsis Campaign Guidelines 2021"
* Age lower than 18

Exclusion Criteria:

* Reason of admission: Cardiac arrest
* Pregnancy
* Abdominal surgery in the past 90 days
* Pre-diagnosis of end-stage renal disease
* History of abdominal trauma
* Body mass index of 30 and above
* Trauma, bleeding or cerebrovascular event that causes increased intracranial pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Change of the Level of Acute Kidney Injury | up to 90 days
  Kidney damage will be monitored according to the KDIGO (Kidney Disease Improving Global Outcomes) classification.
Mortality | at 30th day of admission
  Mortality in first 30 days
Mortality | at 90th day of admission
  Mortality in first 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- UHS Izmir Bozyaka Education and Research Hospital, Izmir, Karabağlar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Leone M, Asfar P, Radermacher P, Vincent JL, Martin C. Optimizing mean arterial pressure in septic shock: a critical reappraisal of the literature. Crit Care. 2015 Mar 10;19(1):101. doi: 10.1186/s13054-015-0794-z. PMID 25888071
- [Background] Silva S, Teboul JL. Defining the adequate arterial pressure target during septic shock: not a 'micro' issue but the microcirculation can help. Crit Care. 2011;15(6):1004. doi: 10.1186/cc10486. Epub 2011 Nov 2. PMID 22047945
- [Derived] Ozkarakas H, Tekgul ZT, Arslan M, Bilgin MU, Eker HE, Okur O, Calik B. Does Maintaining a Targeted Abdominal Perfusion Pressure Reduce Renal Damage in Patients with Septic Shock?: A Randomized, Controlled, and Open-label Study. Balkan Med J. 2023 Oct 20;40(6):415-421. doi: 10.4274/balkanmedj.galenos.2023.2023-5-9. Epub 2023 Sep 18. PMID 37721127